CLINICAL TRIAL: NCT02958605
Title: Smartphone Medical Applications to Reduce Treatment Dosage Errors in Pediatric Resuscitation; a Randomized Simulation Trial
Brief Title: Smartphone Apps for Pediatric Resuscitation
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Medical Protective Association (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, Principal investigator, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SMARTER1
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Status Epilepticus; Anaphylaxis
Keywords: Children; resuscitation; smartphone
MeSH Terms: conditions — Status Epilepticus; Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone (Experimental): Smartphone application
  Interventions: Device: Smartphone apps
- Handbook (Experimental): Resuscitation handbook who provides drug dosages for each weight for children. For example, at the page of 15 kg, it is written that the dosage of epinephrin is 1.5 cc of 1: 10 000.
  Interventions: Device: Handbook

INTERVENTIONS:
Device: Smartphone apps — If already own a smartphone application dedicated to calculate medication dosage for children, the participant will be allowed to use his/her own application. Otherwise, the resident will be offered to chose among a list of applications paid by the research team (PediSafe, PediStat, Palm Pedi, Safedose, EZdrip peds). He/she will be instructed to practice with a few time at home before doing the simulations.
  Arms: Smartphone
Device: Handbook — Resuscitation handbook who provides drug dosages for each weight for children. For example, at the page of 15 kg, it is written that the dosage of epinephrin is 1.5 cc of 1: 10 000.
  Arms: Handbook

SUMMARY:
Medication errors are common in children. Characteristics of errors during critical situations in the Emergency Department are ill-defined and might be more frequent than previously thought. However, optimal strategies to eliminate the risk of prescribing errors remain unknown.

Many smartphone apps have been suggested over the last years with some of them designed to calculate medication dosage for children. The impact of these apps to decrease dosage error has never been evaluated in resuscitation setting.

The aim of the study is to evaluate whether the use of a smartphone application designed to calculate medication doses decreases prescribing errors among residents during pediatric simulated resuscitations.

This will be a crossover-randomized trial using high fidelity simulation among 40 residents rotating in the pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Residents (PGY1 to PGY4)
* Completing a rotation in pediatric emergency

Exclusion Criteria:

* Residents who previously participated in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Medication error | During resuscitation
  The primary outcome is the presence of a medication error. An error will be defined as a drug dose varying by more than 20% from the recommended dose or by incorrect route.

SECONDARY OUTCOMES:
Proportion of tenfold error | During resuscitation
  A tenfold error will be defined as a drug dose varying by a factor of 10 compared to the recommended dose.
Time for prescribing the first medication | During the simulation (10 minutes)
  Time from the beginning of the simulation and complete prescription (oral or written) of the first medication.
Error in bolus medication | during simulation
  An error in bolus medication will be defined as a drug dose varying by more than 20% from the recommended dose or by incorrect route.
Error in perfusion medication | during simulation
  An error in perfusion medication will be defined as a drug dose varying by more than 20% from the recommended dose. This can be related to a preparation error or a flow error.
User satisfaction | 2 weeks
  Satisfaction of the resident with both tools using a Visual analog scale
User confidence | 2 weeks
  Confidence of the resident while using both tools using a Visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No